CLINICAL TRIAL: NCT04707027
Title: Interval of Disease Inactivity After Complete Polypoidal Regression on ICGA in Eyes With Polypoidal Choroidal Vasculopathy Following Intravitreous Aflibercept Treatment
Brief Title: Interval of Disease Inactivity After Complete Polypoidal Regression in PCV Receiving Aflibercept
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Voraporn Chaikitmongkol, Assistant Professor, Chiang Mai University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OPT-2563-07160
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — aflibercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complete polypoidal regression arm (Sham Comparator): follow up monthly with color fundus photography and OCT at each visit
  Interventions: Other: Defer treatment
- incomplete polypoidal regression arm (Active Comparator): continue treatment with aflibercept injection (treat and extend regimen)
  Interventions: Drug: Aflibercept Injection (2 mg/0.05 ml)

INTERVENTIONS:
Drug: Aflibercept Injection (2 mg/0.05 ml) — Intravitreal aflibercept injections (treat and extend regimen)
  Other Names: Eylea
  Arms: incomplete polypoidal regression arm
Other: Defer treatment — Follow up with fundus photo and OCT every 4 weeks
  Arms: complete polypoidal regression arm

SUMMARY:
Polypoidal choroidal vasculopathy (PCV), a subtype of neovascular age-related macular degeneration (NV AMD), is an important cause of central visual loss, especially among Asian and African descendants. PCV is characterized by the presence of hyperfluorescent polypoidal lesions, with or without branching vascular network, identified on indocyanine green angiography (ICGA), currently the gold standard for PCV diagnosis.

In addition to visual improvement from baseline, polypoidal regression or complete disappearance of polypoidal lesions on ICGA has been considered an important treatment outcome in large PCV trials including the PLANET1 and EVEREST II2 studies. Rate of polypoidal regression following intravitreous aflibercept monotherapy was 33% in the PLANET study1 year 2 and ranged between 55% to 78% in other Asian cohorts.3-4

Recently, our previous investigation5 on the timing of polypoidal regression following a fixed-dosing aflibercept monotherapy (3 initial monthly injections, then q 8 weeks until 1 year) in 40 Thai PCV eyes suggested that, among 22 eyes (55%) with polypoidal regression at 1 year, a majority of them showed complete polypoidal regression before 6 months (median duration of complete regression: 3 months (IQR, 2 months to 6 months).

However, due to the fixed-dosing regimen used in previous study, there are limited data on how often polypoidal lesions remain regressed on ICGA when the treatment is deferred in eyes with polypoidal regression, nor what changes might be seen subsequently on OCT when treatment is deferred in this situation. Therefore, this study aims to determine the changes seen on OCT subsequent to complete regression of polypoidal lesions on ICGA in PCV eyes following intravitreous aflibercept treatment.

Results from this study may provide some insights on longer-term PCV management

DETAILED DESCRIPTION:
Primary objective:

To determine how long there is CNV inactivity on OCT (absence of intraretinal thickening, intraretinal cystoid abnormalities, subretinal fluid, or enlarging pigment epithelial detachments) in eyes with complete polypoidal regression on ICGA after receiving intravitreous aflibercept injections over 2 years for PCV

Secondary objectives:

1. To determine the rate of polypoidal regression compared with baseline at 3, 6, 12, and 24 months following intravitreous aflibercept "treat and extend" regimen
2. To determine the visual acuity change from baseline to 1 and 2 years following intravitreous aflibercept "modified treat and extend" regimen and its correlation with OCT or ICGA activity.
3. To determine the correlation of changes at week 12 with changes at 12 months and 24 months
4. To determine the incidence of newly developed or recurrent polypoidal lesions in eyes with complete polypoidal regression after aflibercept treatment "treat and extend" regimen over 2 years

Study design:

Multi-center prospective case series. The overall study duration will be 3 years; 1 year for recruitment and 2-year follow-up for each participant

Methods

* Overall study duration for each participant will be 24 months
* Eligible participants will receive 3 initial monthly intravitreous 2-mg aflibercept injections (week 0, 4, 8), then management will be based on ICGA findings at week 12 as follows:
* Complete polypoidal regression on ICGA: defer intravitreous aflibercept injection, and follow-up monthly with OCT monitoring thereafter until 1 year, and bimonthly in year 2. If subretinal or intraretinal fluid is seen on OCT during the follow-up period, an interval of disease inactivity is determined. Such study eye with re-activation is considered met primary end point and will receive intravitreous anti-VEGF treatment according to "treat and extend" regimen as described below.
* Incomplete or worsening polypoidal regression on ICGA: continue additional 3 intravitreous aflibercept injection, and repeat ICGA at week 24

  * At week 24, if there is a presence of complete polypoidal regression on ICGA, defer intravitreous aflibercept injection, and follow-up monthly with OCT monitoring thereafter until 1 year, and bimonthly in year 2. If subretinal or intraretinal fluid is seen on OCT during the follow-up period, an interval of disease inactivity (primary outcome) is determined. Such study eye with re-activation is considered met primary end point and will receive intravitreous anti-VEGF treatment according to "treat and extend" regimen as described below.
  * At week 24, if there is partial or no regression of polypoidal lesion, continue intravitreous aflibercept injection with "treat and extend" regimen, which the follow-up interval can be extended by 4 weeks up to 16 weeks if no disease activity identified on color fundus photography or OCT. If disease activity recurs, shorten follow-up interval by 4 weeks, remain injections at that interval until fluid resolved, and re-extend by 2 weeks. Treatment interval will not be less frequent than every 4 weeks (according to an approved label of intravitreous aflibercept in Thailand). During follow-up, if an investigator suspect the presence of complete polypoidal regression based on OCT findings, ICGA can be performed at any visit. If complete polypoidal regression is present, defer the treatment and follow-up monthly with OCT monitoring in year 1, and bimonthly in year 2.
  * Photodynamic therapy can be applied at 1 year, if persistent fluid on OCT is identified despite continuous intravitreous aflibercept injections.

Investigations at each visit

* Visual acuity measurement, color fundus photography (CFP), and SD-OCT will be performed at each visit
* Fundus fluorescein angiography (FA) and indocyanine green angiography (ICGA) will be performed at week 0 (baseline), 3, 6, 12, and 24 months, and at any time point showing a recurrence of disease activity in eye that previously shown complete polypoidal regression on ICGA, or at any time point an investigator suspect the presence of complete polypoidal regression based on OCT findings.

Definitions:

* Disease activity on color fundus photography is defined as a presence of new retinal or subretinal or sub-RPE hemorrhage
* Disease activity on OCT is defined as a presence of intraretinal or subretinal fluid or new pigment epithelial detachment
* Polypoidal regression is defined as complete absence of hyperfluorescent lesions in an area that previously had a polypoidal lesion on ICGA at baseline
* Partial polypoidal regression is defined as decrease of hyperfluorescent polypoidal lesions either in size or number or both in an area previously identified as a polypoidal lesion on ICGA at baseline
* Persistent or worsening polypoidal regression is defined as a persistent or enlargement in size and number of hyperfluorescent lesions in an area previously identified as a polypoidal lesion on ICGA at baseline
* Newly developed polypoidal lesion is defined as a presence of a polypoidal lesion not previously identified on ICGA at baseline
* Recurrent polypoidal lesion is defined as a polypoidal lesion in an area previously identified as polypoidal regression on ICGA.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥18 years
* Diagnosis of treatment-naïve PCV in either eye

  * PCV is defined according to the following criteria Presence of focal subretinal ICGA hyperfluorescence within the first 6 minutes, plus one of the followings; 1) subretinal orange nodule corresponds to hyperfluorescent nodule on ICGA, 2) massive submacular hemorrhage of 4 disc area or larger, 3) nodular appearance on stereoscopic viewing, 4) pulsatile polypoidal lesion, 5) abnormal vascular channel supplying the polypoidal lesion, 6) hypofluorescent halo around the nodule6
* If any participant presents with bilateral PCV in which both eyes are eligible for the study, the eye with worse vision will be chosen as the study eye

Exclusion Criteria:

* Presence of co-existing vision threatening conditions in the study eye, e.g., diabetic retinopathy, or retinal vascular occlusion
* Presence of ocular or periocular infections, active intraocular inflammation, or known hypersensitivity to aflibercept or any of the excipients in aflibercept
* Inability to obtain good quality imaging due to ocular media abnormalities
* Contraindicate for FFA or ICGA due to the following conditions:

  * Allergic to fluorescein or indocyanine green dye
  * Allergic to iodine or seafood
  * Impaired kidney or liver functions
* Not able to follow up according to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Interval of disease activity on color fundus photography or optical coherence tomography | 1 to 24 months
  * Disease inactivity on color fundus photography is defined as an absence of new retinal or subretinal or sub-RPE hemorrhage on color fundus photography compared with baseline
  * Disease inactivity on OCT is defined as an absence of intraretinal thickening or CME or subretinal fluid or PED or enlarging PED on OCT

OTHER OUTCOMES:
Systemic adverse event | 1 to 24 months from baseline
  incidence of stroke or myocardial infarction
Ocular adverse event | 1 to 24 months from baseline
  incidence of post-injection endophthalmitis, retinal detachment, or vitreous hemorrhage, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Voraporn Chaikitmongkol, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No